CLINICAL TRIAL: NCT02668159
Title: Cardiometabolic Health Effects and Mechanisms of Action of Fish Nutrients
Brief Title: Pilot Study on Metabolic Effects of Fish Peptides and Vitamin D
Acronym: BONITO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie-Claude Vohl, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BONITO 2015-090
Record Dates: First submitted 2015-09-01; First posted 2016-01-29 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Prediabetes; Insulin Resistance
MeSH Terms: conditions — Prediabetic State; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fish peptide (Experimental)
  Interventions: Dietary Supplement: Fish peptide supplement
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: Vitamin D supplement
- Fish peptide + Vitamin D (Experimental)
  Interventions: Dietary Supplement: Fish peptide + Vitamin D3 supplements
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish peptide supplement — 6 capsules of fish peptide supplement (3g/each) administered prior to one of the OGTT
  Arms: Fish peptide
Dietary Supplement: Vitamin D supplement — 1 tablet of vitamin D3 (1000 UI) administered prior to one of the OGTT
  Arms: Vitamin D
Dietary Supplement: Fish peptide + Vitamin D3 supplements — 6 capsules of fish peptide (3g/each) + 1 tablet of vitamin D3 (1000 UI) administered prior to one of the OGTT
  Arms: Fish peptide + Vitamin D
Dietary Supplement: Placebo — 7 tablets of placebos administered prior to one the OGTT
  Arms: Control

SUMMARY:
The overall goal of this study is to investigate the effects and the mechanisms of action of a fish peptide and vitamin D on glucose metabolism, insulin secretion, and cardiometabolic risk profile in overweight men. Transcriptomic and metabolomic approaches will be used to study the acute physiological effects of fish nutrients and to discover gene/metabolite networks that underlie these effects.

DETAILED DESCRIPTION:
Sedentary lifestyle and excess calorie intake have contributed to a dramatic increase in the occurrence of obesity, metabolic syndrome (MetS), type 2 diabetes (T2D) and cardiovascular disease (CVD) The first step in reducing the excessive CVD risk associated with the presence of the MetS is the adoption of a healthier lifestyle. A balanced diet, including high-nutritive and low-energy foods such as fish, is an important component of a healthy diet. Fish is a major source of n-3 PUFA, high-quality protein, and other essential nutrients such as vitamin D. Fish consumption may therefore improve the components of the MetS and reduce the incidence of T2D and CVD in obese subjects.The foundation of this project stems from the well-recognized fact that few Canadians meet the weekly dietary recommendation for fish consumption (i.e. 2 servings/week) and thus intakes of both n-3 polyunsaturated fatty acid (PUFA) and fish protein are low in the general population, and even lower in obese subjects. Since some people simply dislike fish and because certain types of fish contain toxic contaminants, including heavy metals and environmental pollutants, fish consumption remains low. Therefore, dietary choices limit intake of its key nutrients, thus increasing risk for MetS, T2D and CVD. Also, fish is one of the richest food sources of dietary vitamin D which may also contribute to the health benefits of fish consumption. Indeed, it is currently estimated that ∼40% of Canadians have low serum 25-hydroxyvitamin D [25(OH)D] concentrations (≤50 nM) and that ∼70% are below 75 nM. In addition, obesity is an important risk factor for low serum 25(OH)D.The main objective of this study is to investigate the acute effects and mechanisms of action of fish peptide and vitamin D on glucose metabolism, parameters of insulin sensibility and secretion, and cardiometabolic risk profile in overweight men.

A four-arm randomized crossover design will be used to test the metabolic effects of consuming prior to a 3h-oral glucose tolerance test (OGTT), supplements containing either fish peptide (3 grams), vitamin D3 (1000 IU), a combination of fish peptide + vitamin D3 or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI 25-40 kg/m2)
* fasting triglycerides ≥ 1.5 mmol/L
* fasting insulin ≥ 60 pmol/L
* non-smoking
* stable weight in the past 3 months

Exclusion Criteria:

* diabetes
* chronic diseases
* taking drugs that could affect glucose or lipid metabolism
* taking dietary supplements or natural health products
* major surgery 3 months prior to the study
* fish or seafood allergy
* lactose intolerance

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum glucose area under the curve (Glucose AUC) | 0-180 min
  The area under the curve for serum glucose concentration is calculated from 0-180min after 75g glucose is ingested

SECONDARY OUTCOMES:
Serum insulin area under the curve (Insulin AUC) | 0-180 min
  Area under the curve for serum insulin
Serum C-peptide area under the curve (C-peptide AUC) | 0-180 min
  Area under the curve for serum C-peptide
Serum triglycerides concentrations | -15, 0, 15, 30, 60, 120, 180 min post 75g glucose
  changes in the triglycerides concentration at each time point of the OGTT
Serum 25(OH)D concentrations | 4 weeks
  Changes in the 25(OH)D concentration measured before each OGTT
Cardiometabolic risk profile in serum | 4 weeks
  Changes in cardiometabolic profile measured in serum before each OGTT
Gene expression profile | 4 weeks
  peripheral blood mononuclear cells (PBMCs) gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Vohl, Principal Investigator — Instute of Nutrition and Functional Foods, Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Laval University, Québec, Canada